CLINICAL TRIAL: NCT02962882
Title: A Multi-Centre, Open, Non-controlled, Clinical Investigation to Evaluate the User Friendliness and Wear Time of Multi-layer Foam Dressings With Safetac® for Pressure Injury Prevention in the Intensive Care Unit
Brief Title: Pressure Injury Prevention in the ICU With Multi-Layer Foam Dressings
Acronym: PUP16_01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUP16_01
Record Dates: First submitted 2016-08-23; First posted 2016-11-15 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Pressure Incidence Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. Mepilex Border Sacrum (Safetac) (Experimental): A dressing that is a flexible, self-adherent, profylactic, absorbent pad in three layers to be used on the sacrum area at pressure points in patients in the ICU, prone to get pressure injuries (PI).
  Interventions: Device: Mepilex Border
- B. Mepilex Border Heel (Safetac) (Experimental): A dressing that is a flexible, self-adherent, profylactic, absorbent pad in three layers to be used on the heels (on both left and right heels), in patients in the ICU, prone to get pressure injuries (PI).
  Interventions: Device: Mepilex Border

INTERVENTIONS:
Device: Mepilex Border — Multi-layer Foam Dressings

SUMMARY:
A Multi-Centre, Open, Non-controlled, Clinical Investigation to Evaluate the User Friendliness and Wear Time of Multi-layer Foam Dressings With Safetac® for Pressure Injury Prevention in the Intensive Care Unit

DETAILED DESCRIPTION:
This was a multi-centre, open, non-comparative, prospective, clinical investigation involving 50 enrolled subjects using competitive enrolment at two sites in the United States of America (USA). The study was conducted on subjects at risk of developing PIs according to investigators' judgment and facility protocol being treated in ICUs. The target subjects were male and female, 18 years and above, with an expected hospital stay of 4-6 days. An evaluable subject was defined as a subject that was enrolled and had data for at least one visit after the baseline visit. There were two parts to the study: Part A: Mepilex Border/Protect Sacrum; Part B: Mepilex Border/Protect Heel (on both left and right heels), used within intended use and according to IFU.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at risk for developing a pressure injury to the heels and/or sacrum
* Aged ≥ 18 years
* Patient or his/her legal representative is able to understand and voluntarily sign the informed consent
* Estimated treatment period in ICU for patient at least 4-6 days

Exclusion Criteria:

* Patient has a pressure injury or blistering on sacrum and/or heels
* Patient with known or suspected sensitivity to any of the components of the products being evaluated
* Patient included in other clinical investigations at present or within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Potter, BSN, RN, Principal Investigator — AnMed Health Medical Center
Locations (2):
- United States (2):
  - Anmed Health, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigation period: Sept 2016 - Nov 2016. This study was conducted in two sites in the US, on patients being treated in an ICU who were at risk of developing pressure injuries.
  The target subjects were male or female, aged 18 years or above, with an expected stay of 4-6 days in an ICU.
Groups:
- Mepilex Border Dressing All: A dressing that is a flexible, self-adherent, profylactic, absorbent pad in three layers to be used on the sacrum area and heels at pressure points in patients in the ICU, prone to get pressure injuries (PI).
  Mepilex Border: Multi-layer Foam Dressings
Period: Overall Study
Arm/Group | Mepilex Border Dressing All
Started | 50
Completed | 14
Not Completed | 36
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Transfer from ICU | 32

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Mepilex Border Dressing Heel and Sacrum Together: A dressing that is a flexible, self-adherent, profylactic, absorbent pad in three layers to be used on the sacrum area and heels at pressure points in patients in the ICU, prone to get pressure injuries (PI).
  Mepilex Border: Multi-layer Foam Dressings
Arm/Group | Mepilex Border Dressing Heel and Sacrum Together
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: User Friendliness of Both Sacrum and Heel (Left & Right) Dressings: Comfort, Conformability, Acceptability, the Handling at Application and Ease of Inspection of the Dressings as Well as Reapplication
Description: User friendliness judged by site staff, with the following variables; Ability to stay in place Facilitation of inspection Ease of reapplication Conformability to the body Overall impression of dressing
  *NOTE: Since subjects typically left the ICU earlier than expected (the study protocol stipulated that the test dressing should be left in place for 3 days or longer, however typically the subjects left the ICU department after one day), not all subjects completed the full study period/all study visits.
  Furthermore, since not all assessment visits were completed for each subject or a dressing change was not required, the total number of all visits exceeds the total number for each variable. This was because the subject did not undergo a dressing application/removal or that the question was not relevant at a given visit (some questions were only relevant for dressing applications, some questions were only relevant for dressing removals or only relevant for dressing inspections).
Time Frame: 4-6 days
Population: ITT population As a dressing change was not required at all visits, the total number of dressing changes evaluated vary for each variable and a question was perhaps not relevant at a given visit (some questions were only relevant for dressing applications, some were only relevant for dressing removals or only relevant for dressing inspections).
Measure: Count of Units; unit: Dressing changes evaluated
Units Other Than Participants: Dressing changes evaluated
Groups:
- Mepilex Border Dressing Heel; Mepilex Border Dressing Sacrum: A dressing that is a flexible, self-adherent, profylactic, absorbent pad in three layers to be used on the sacrum area and heels at pressure points in patients in the ICU, prone to get pressure injuries (PI).
  Mepilex Border: Multi-layer Foam Dressings
Arm/Group | Mepilex Border Dressing Heel | Mepilex Border Dressing Sacrum
Number analyzed (Participants) | 50 | 50
Number analyzed (Dressing changes evaluated) | 119 | 128
Dressing changes evaluated
  Ease/speed of application of dressing: number analyzed (Dressing changes evaluated) | 87 | 94
  Ease/speed of application of dressing: Very Poor | 1 | 1
  Ease/speed of application of dressing: Poor | 6 | 0
  Ease/speed of application of dressing: Good | 14 | 16
  Ease/speed of application of dressing: Very Good | 26 | 28
  Ease/speed of application of dressing: Excellent | 40 | 49
  Ease/speed of correct positioning: number analyzed (Dressing changes evaluated) | 87 | 92
  Ease/speed of correct positioning: Very Poor | 0 | 0
  Ease/speed of correct positioning: Poor | 8 | 0
  Ease/speed of correct positioning: Good | 14 | 16
  Ease/speed of correct positioning: Very Good | 26 | 29
  Ease/speed of correct positioning: Excellent | 39 | 47
  Non-adherence to skin at removal: number analyzed (Dressing changes evaluated) | 64 | 73
  Non-adherence to skin at removal: Very Poor | 6 | 1
  Non-adherence to skin at removal: Poor | 6 | 1
  Non-adherence to skin at removal: Good | 17 | 18
  Non-adherence to skin at removal: Very Good | 14 | 24
  Non-adherence to skin at removal: Excellent | 21 | 29
  Ability to stay in place: number analyzed (Dressing changes evaluated) | 85 | 91
  Ability to stay in place: Very Poor | 4 | 0
  Ability to stay in place: Poor | 9 | 4
  Ability to stay in place: Good | 18 | 14
  Ability to stay in place: Very Good | 20 | 29
  Ability to stay in place: Excellent | 34 | 44
  Ability to conform to body contours: number analyzed (Dressing changes evaluated) | 119 | 127
  Ability to conform to body contours: Very Poor | 5 | 1
  Ability to conform to body contours: Poor | 11 | 2
  Ability to conform to body contours: Good | 22 | 26
  Ability to conform to body contours: Very Good | 28 | 32
  Ability to conform to body contours: Excellent | 53 | 66
  Coverage of bony prominence: number analyzed (Dressing changes evaluated) | 119 | 127
  Coverage of bony prominence: Very Poor | 3 | 1
  Coverage of bony prominence: Poor | 8 | 1
  Coverage of bony prominence: Good | 22 | 25
  Coverage of bony prominence: Very Good | 32 | 33
  Coverage of bony prominence: Excellent | 54 | 67
  Ease of removal of dressing: number analyzed (Dressing changes evaluated) | 67 | 75
  Ease of removal of dressing: Very Poor | 4 | 2
  Ease of removal of dressing: Poor | 7 | 0
  Ease of removal of dressing: Good | 20 | 22
  Ease of removal of dressing: Very Good | 13 | 20
  Ease of removal of dressing: Excellent | 23 | 31
  Overall experience: number analyzed (Dressing changes evaluated) | 118 | 128
  Overall experience: Very Poor | 4 | 1
  Overall experience: Poor | 14 | 1
  Overall experience: Good | 21 | 27
  Overall experience: Very Good | 29 | 38
  Overall experience: Excellent | 50 | 61
  Ability to conform to the gluteal cleft: number analyzed (Dressing changes evaluated) | 0 | 126
  Ability to conform to the gluteal cleft: Very Poor |  | 1
  Ability to conform to the gluteal cleft: Poor |  | 2
  Ability to conform to the gluteal cleft: Good |  | 26
  Ability to conform to the gluteal cleft: Very Good |  | 35
  Ability to conform to the gluteal cleft: Excellent |  | 62

2. Primary Outcome: User Friendliness of Both Sacrum and Heel (Left & Right) Dressings: Comfort, Conformability, Acceptability, the Handling at Application and Ease of Inspection of the Dressings as Well as Reapplication
Description: User friendliness judged by site staff, with the following variables; How do you prefer this dressing to your current dressing?
  *NOTE: Since subjects typically left the ICU earlier than expected (the study protocol stipulated that the test dressing should be left in place for 3 days or longer, however typically the subjects left the ICU department after one day), not all subjects completed the full study period/all study visits.
  Furthermore, since not all assessment visits were completed for each subject or a dressing change was not required, the total number of all visits exceeds the total number for each variable. This was because the subject did not undergo a dressing application/removal or that the question was not relevant at a given visit (some questions were only relevant for dressing applications, some questions were only relevant for dressing removals or only relevant for dressing inspections).
Time Frame: 4-6 days
Population: ITT population As a dressing change was not required at all visits, the total number of dressing changes will vary for each variable and a question was perhaps not relevant at a given visit (some questions were only relevant for dressing applications, some were only relevant for dressing removals or only relevant for dressing inspections).
Measure: Count of Units; unit: Number of dressing changes
Units Other Than Participants: Number of dressing changes
Arm/Group | Mepilex Border Dressing Heel | Mepilex Border Dressing Sacrum
Number analyzed (Participants) | 50 | 50
Number analyzed (Number of dressing changes) | 39 | 58
Number of dressing changes
  Much better than | 6 | 6
  Better than | 16 | 29
  Equal to | 10 | 22
  Not as good as | 7 | 1

3. Secondary Outcome: Wear Time (Days) for First Dressing
Description: Maximum length of wear time/stay on ability of dressings in ICU.
Time Frame: 4-6 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepilex Border Dressing Heel | Mepilex Border Dressing Sacrum
Number analyzed (Participants) | 50 | 50
Participants
  0 Day | 2 | 2
  1 Day | 23 | 23
  2 Days | 17 | 19
  3 Days | 4 | 4
  4 Days | 2 | 2
  5 Days | 2 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 months.
Arm/Group | Mepilex Border Dressing All
All-Cause Mortality (participants affected / at risk) | 4/50
Serious Adverse Events (participants affected / at risk) | 7/50
Other Adverse Events (participants affected / at risk) | 1/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Border Dressing All (N=50)
Death (General disorders) | 4 (4)
Prolongation of existing hospitalization (Infections and infestations) | 2 (2) — Subject developed sepsis related to possible pneumonia on 18Nov2016. Mechanical ventilation weaning and vasopressor medication weaning were delayed, thus prolonging the subject's hospitalization.
Bowel perforation (Gastrointestinal disorders) | 1 (1) — Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Border Dressing All (N=50)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Worsening Sepsis (Infections and infestations) | 1 (1)
Possible pneumonia and sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes